CLINICAL TRIAL: NCT02997540
Title: Evaluation of the Effect of Body Position and Probe Position on the Localization of Breast Mass in Free-Hand Breast Ultrasound Examination
Brief Title: Effect of Body Position and Probe Position on the Localization of Breast Mass
Status: Terminated | Type: Observational
Why Stopped: Successfully obtained sufficient data to complete this research project.
Sponsor: MetriTrack, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BVN G-1000
Record Dates: First submitted 2016-12-07; First posted 2016-12-20 (Estimated); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Breast Diseases
Keywords: female breast lesion; ultrasound examination
MeSH Terms: conditions — Breast Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- female breast ultrasound exam: females with at least one benign or probably benign mass, up to 2 cm in size, in one breast, detected during a standard-of-care breast ultrasound examination

SUMMARY:
The purpose of this study is to demonstrate that BVN G-1000 can precisely and consistently measure the position of female breast lesions regardless of patient rotation and probe angle during ultrasound examination.

DETAILED DESCRIPTION:
The proposed research consists of quantitatively detecting and reporting the effect of body rotation and ultrasound probe position on the breast on the position of breast lesions relative to the breast nipple and body orientation planes, required for positional annotations, in female subjects at one study visit. Measurements will be manually and automatically recorded by two ultrasound operators with each image and will be compared among these conditions to detect effects of probe position and probe orientation and patient's body position relative to the exam table. The manual and automated measurements will be compared to determine the differences between the data obtained using the two different methods.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. 21-70 years of age
3. Known palpable or non-palpable benign or probably benign breast mass or masses, less than 2 cm in maximum diameter and at least 4 cm away from the nipple, from a previous ultrasound examination

Exclusion Criteria:

1. Women with cardiac pacemaker or portable defibrillator
2. Women with known breast cancer or suspicious lesions
3. Pregnant and lactating women
4. Women who have breast implant(s)
5. Women who have had prior breast surgical intervention not including breast needle biopsy, in the same breast with the qualifying target mass.
6. Women with the target finding to be mapped within a distance of 4 cm from patient's nipple.
7. Women with multiple similar qualifying targets in close proximity (less than 4 cm between targets).
8. Women with history of allergy to medical-grade adhesive tape or ultrasound gel
9. Women whose weight is over 250 pounds

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Females of any ethnic group who meet all inclusion and none of the exclusion criteria will be eligible for enrollment
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
movement of a given ultrasound breast lesion | study completion, an average of 1 day
  movement of a given ultrasound breast lesion between different operators and between different body rotation positions and probe positions and orientations

CONTACTS AND LOCATIONS:
Locations (1):
- Evanston Hospital, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided